CLINICAL TRIAL: NCT06795568
Title: Examination of Fertility Awareness with an Integrative Approach: a Mixed-method Multi-centre Research Study
Brief Title: Complex Fertility Awareness Study - Hungary
Acronym: FAIR-HU
Status: Not yet recruiting | Type: Observational
Sponsor: University of Pecs (Other)
Collaborators: University of Debrecen (Other); Dunamenti REK Reproduction Center (Unknown)
Responsible Party: Principal Investigator, Prémusz Viktória, Dr. PRÉMUSZ Viktória Ph.D, University of Pecs
Other Study IDs: BM/30545- 3 /2023; NKFI FK-147404 (Other Grant/Funding Number: National Research, Development and Innovation Office (NRDI Office))
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Infertility, Sterility, Reproductive, Reproductive Sterility, Sterility, Subfertility, Sub-Fertility
Keywords: Fertility; integrative approach; infertility; assisted reproductive techniques, IVF; health behaviour; physical activity; dietary
MeSH Terms: conditions — Infertility; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to investigate integrative fertility awareness and its impact on assisted reproductive techniques (ART) in Hungary. It analyzes fertility awareness, health-movement behavior, physical literacy, dietary patterns, psycho-social distress, socio-demographic parameters, and stress biomarkers across four fertility centers. The study employs a mixed-method approach. The research aims to review and analyze the factors of integrative fertility awareness on the course and outcome measures of assisted reproductive techniques (ART) at different fertility centers in Hungary in a mixed-method study.

DETAILED DESCRIPTION:
Introduction:

The United Nations warns that global demographic trends indicate the world's population is projected to reach 9.7 billion by 2050 and 11 billion by the end of the 21st century. While some countries experience population decline, many are transitioning to an aging population due to longer life expectancy, delayed childbearing, and declining fertility rates. In Hungary, the population has been declining since 1981, with live births remaining below pre-2008 crisis levels. In 2020, there were only 92,000 live births, a 52% decrease compared to 1975.

Hungary's lower birth rate is attributed to infertility, and approximately 10-15% of couples face fertility problems. The World Health Organization (WHO) reports a 12-15% incidence of fertility disorders, with secondary infertility prevalence at 18.0% in Central and Eastern Europe. Due to this in-vitro fertilization (IVF), has increased. Factors affecting IVF outcomes include age, sperm quality, embryo quality, and endometrial thickness. Public policies provide freely available examinations and medicines, emphasizing integrative analysis and add-on treatments to enhance success rates and participant experience. However, no research currently analyzes health behaviors related to reproductive treatments from a fertility awareness perspective.

Significance of Study:

This study is important because previous studies emphasize variations in infertility outcomes related to recreational physical activity (PA). However, the ideal PA metrics (weekly minutes) are not yet defined, and comprehensive investigations considering sleep and awareness are scarce. Hungarian researchers concentrate on psychosocial aspects in infertile couples but have not incorporated lifestyle assessments. Their innovative concept of integrative fertility awareness distinguishes their work globally.

This study will be done in four different centers including; (1) Assisted Reproduction Unit, Department of Obstetrics and Gynaecology, University of Pécs, National Laboratory on Human Reproduction, (2) University of Debrecen, Clinical Center (DEKK), Health Service Units, Center for Assisted Reproduction, (3) Róbert Károly Infertility Center, Dunamenti REK Infertility Centre, (4) Buda Infertility Center, Dunamenti REK Infertility Centre.

All female patients with both female and male factors of infertility who were indicated for fertility treatment (IVF/ICSI) and their spouses will be consecutively invited to participate in the study.

Objectives:

Some of the objectives to be answered through this proposal are:

Objective 1: Investigation of fertility awareness (reproductive health literacy, fertility awareness, fertility treatment compliance) of female patients with infertility diagnoses and indicated for fertility treatment (Pre-ART/ART) by socio-demographic parameters, Objective 2: Mapping of physical activity patterns with subjective and objective measurement methods based on the 24h health-movement behavior concept (amount and intensity of physical activity - sedentary behavior - sleep quality and quantity) and physical literacy.

Objective 3: Investigating the relationship between dietary patterns (with special regard to non-prescription supplements and fertility awareness.

Methods:

The study will collect socio-demographic information through questions about age, education level, income, marital status, partnership duration, infertility duration, BMI, and lifestyle habits. For the assessment of physical activity (PA), sedentary behavior, and sleep, participants will self-report their exercise habits using a PA diary and the survey method. Participants' self-reported PA will be compared with objective measures collected using Triaxial ActiGraph GT3X+ accelerometers. These accelerometers, along with ActiLife 6 software, have high sensitivity (over 98%) and specificity (over 99%). Discrepancies between objective and self-reported PA emphasize the need to improve physical literacy among those undergoing assisted reproductive technology (ART) treatment. We plan to assess it using a Physical Literacy Questionnaire.

In additional, the fertility awareness assessment will be done by use of a modified version of the Fertility-Awareness Questionnaire (FAQ). On dietary supplements, the study will investigate dietary patterns and non-prescription supplements based on self-reports from respondents. For, laboratory measures in our study, we'll measure oxidative stress markers using the ELISA method. Energy balance will be exeminde with CGMs.

The statistical analyses will be conducted using IBM SPSS Statistics 27.0 for Mac. Methods include the Kolmogorov-Smirnov test for data distribution, the Mann-Whitney U-test for continuous variables, Spearman's rank correlation for associations, and multivariate linear regression for predicting outcomes. Logistic regression evaluates covariate effects on live births. Posthoc power analysis will use G*Power software. Data will be expressed as mean ± SD and medians with 25th and 75th percentiles, with significance at p˂0.05. The dataset supporting the conclusions of this article will be available from the repository of the University of Pécs (PEA, https://pea.lib.pte.hu/)

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will be BMI ≥ 18 kg/m2 and ≤ 38 kg/m2, 18 to 45 years of age, having undergone not more than three unsuccessful cycles and no significant health risk relevant to the ART procedure and outcome (metabolic and vascular diseases including diabetes mellitus, metabolic syndrome, fatty liver diseases and atherosclerosis

Exclusion Criteria:

* Participants diagnosed with any mental disorders and significant physical or mobility impairments will be excluded.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All female patients with both female and male factors of infertility who were indicated for fertility treatment (IVF/ICSI) will be randomly enrolled to participate in the study. Spouses will be enrolled based on the above invitation.
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Level of Fertility Awareness | 18 month
  The level of fertility awareness measured by Fertility Awareness Survey (FAS and FAS-M) questionnaire. The Hungarian version of the Fertility Awareness Survey (FAS) will be used to evaluate knowledge and attitudes regarding assisted reproductive technologies (ART). Originally developed by Daniluk et al., the FAS includes separate knowledge sections for women and men. The questionnaire has three sections: self-assessed knowledge and attitudes toward ART, factual knowledge about general fertility, and ART-related knowledge. Participants will indicate their knowledge and attitudes, and respond to statements about fertility and ART.
Primary outcome of the MART - Live birth | 18 month
  Live birth with a gestational age of ≥ 20 weeks, reflecting the World Health Organization definition.

SECONDARY OUTCOMES:
Fertility-Related Stress and Coping (COMPI FPSS & CSS) | 18 month
  The Copenhagen Multi-Centre Psychosocial Infertility Study (COMPI) Fertility Problem Stress Scale (FPSS) and Coping Strategy Scale (CSS) are widely used to measure infertility-related stress and coping mechanisms. The FPSS assesses stress across domains like personal, social, and partner-related dimensions, while the CSS evaluates strategies such as active avoidance, seeking support, or problem-solving. These tools have been extensively validated in diverse populations (Schmidt et al., 2003; 2005), providing insights into the psychological burden of infertility and coping efficacy.
Screening of Emotional Maladjustment (SCREENIVF) | 18 month
  SCREENIVF is a screening tool designed to identify emotional maladjustment in individuals undergoing fertility treatment. It assesses dimensions such as anxiety, depression, and perceived control, offering a quick yet reliable way to detect individuals at risk of emotional distress. Its development (Verhaak et al., 2010) ensures its applicability in fertility care settings, promoting early interventions to support mental health.
Sexual Life (Fertility Problem Inventory - Sexual Concerns Subscale, FPI-S) | 18 month
  The Fertility Problem Inventory (FPI) is a multidimensional measure of the psychosocial impact of infertility, with the Sexual Concerns Subscale (FPI-S) specifically focusing on how infertility affects sexual life. This subscale addresses issues such as sexual satisfaction, intimacy, and the emotional toll of fertility challenges on sexual relationships (Newton et al., 1999).
Mental Health (BDI-9 H and GHQ-12) | 18 month
  The Beck Depression Inventory - Short Form (BDI-9 H) is a shortened version of the BDI, designed to measure depressive symptoms in clinical and non-clinical populations (Beck et al., 1961; Beck & Steer, 1984). It is widely used in studies involving individuals experiencing fertility-related distress.
  The General Health Questionnaire (GHQ-12) is a brief, reliable tool to screen for general mental health issues, including anxiety and depression. Its adaptability and ease of use make it suitable for assessing overall psychological well-being in fertility-related contexts (Goldberg & Williams, 1988).
Quality of Life (FertiQoL and WHOQoL-BREF) | 18 month
  The Fertility-Related Quality of Life Questionnaire (FertiQoL) is a comprehensive tool designed to measure the impact of fertility problems on quality of life. Developed by Boivin et al. (2011) in collaboration with the World Health Organization, it evaluates four core domains: emotional, mind-body, relational, and social. It also includes optional treatment and core modules. The FertiQoL is extensively validated and widely used in fertility research, providing insights into the psychosocial challenges of individuals or couples undergoing infertility treatment. Its multidimensional approach ensures that various aspects of quality of life specific to infertility are captured.
  The WHOQoL-BREF, developed by the World Health Organization, is a shortened version of the WHOQoL-100. It evaluates quality of life across four key domains: physical health, psychological health, social relationships, and environment. This 26-item questionnaire is validat
Self-reported physical activity and sleep (GPAQ, PAHCO-12 and AIS) | 18 month
  The 24h HMB combines PA and sleep. The Global Physical Activity Questionnaire (GPAQ), developed by the World Health Organization (WHO), is a widely used tool for assessing physical activity in different domains: work, transportation, and leisure time. It captures information about intensity, duration, and frequency of physical activity, as well as sedentary behavior (Armstrong & Bull, 2006).
  The Physical Activity-Related Health Competence (PAHCO-12) is a concise instrument for assessing an individual's competence in health-related physical activity. It evaluates three core dimensions: knowledge about physical activity and its health effects, self-regulation abilities, and intrinsic The Athens Insomnia Scale (AIS) assess insomnia based on ICD-10 criteria. It measures sleep difficulty through eight items covering aspects such as sleep induction, awakenings, sleep duration, and overall quality.
Patient Self-Tracking on PA and energy balance | 18 month
  Examining PA and energy balance on ways that patients will engage with self-tracking activities using mobile apps and ActiGraphGT3Xbt and CareSense CGM.
Complementary medicine (I-CAM-Q) | 18 month
  Complementary Medicine refers to health practices and treatments that are used alongside conventional medical treatments. It includes a broad range of practices, such as acupuncture, herbal medicine, chiropractic care, and others, which aim to improve health and well-being (Ernst, 2005). The I-CAM-Q (International Complementary and Alternative Medicine Questionnaire) is a tool designed to assess individuals' use and attitudes toward complementary and alternative medicine (CAM). It helps in gathering data about CAM use across different populations, offering insights into its prevalence, effectiveness, and integration with conventional care (Cummings & Finnegan, 2017).
Nutritional Supplements in IVF | 18 month
  Self-report on nutritional supplements taken
Health Attitudes and Health Literacy (SHTE and BRIEF) | 18 month
  The Short Health and Treatment Evaluation (SHTE) is a concise questionnaire designed to assess attitudes toward health and treatment. It evaluates individuals' beliefs, perceptions, and readiness to engage in health-related behaviors or interventions. The SHTE is often used in healthcare settings to better understand patient perspectives and improve adherence to treatments.
  The Brief Health Literacy Screening Tool (BRIEF) is a short, validated questionnaire that measures an individual's ability to understand, access, and use health information. It includes simple, direct questions about confidence in filling out medical forms, understanding health information, and seeking help when needed. The BRIEF is widely used for quick assessment in clinical and public health research to identify individuals who may require additional support (Sørensen, K., et al. 2012).
Secondary outcome of the MART - Live birth | 18 month
  Number of oocytes, embryos, chemical pregnancy, clinical pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Viktória Prémusz, PhD, Principal Investigator — University of Pecs; Ákos Várnagy, PhD, Study Director — University of Pecs

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Cross-cultural adaptation and validation of the Global Physical Activity Questionnaire among healthy Hungarian adults. — http://doi.org/10.1186/s12889-020-08477-z
- See also: Oxidative stress in relation to diet and physical activity among premenopausal women — http://doi.org/10.1007/s10389-006-0024-x
- See also: Validity of the Global Physical Activity Questionnaire (GPAQ) in assessing levels and change in moderate-vigorous physical activity and sedentary behaviour — http://doi.org/10.1186/1471-2458-14-1255
- See also: Effects of gender roles, child wish motives, subjective well-being, and marital adjustment on infertility-related stress: a preliminary study with a Hungarian sample of involuntary childless men and women — http://doi.org/10.1007/s00404-013-2835-7
- See also: G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences — http://doi.org/10.3758/bf03193146
- See also: Holistic physical exercise training improves physical literacy among physically inactive adults: a pilot intervention study — http://doi.org/10.1186/s12889-019-6719-z
- See also: Párkapcsolati változások, termékenységi trendek. In S. I. Kolosi Tamás, Tóth István György (Ed.) — http://tarki.hu/sites/default/files/2020-10/146_170_Kapitany_Murinko_web.pdf
- See also: National, regional, and global trends in infertility prevalence since 1990 — http://doi.org/10.1371/journal.pmed.1001356
- See also: Plasma, urinary, and salivary 8-epi-prostaglandin f2alpha levels in normotensive and preeclamptic pregnancies — http://doi.org/10.1067/mob.2000.108877
- See also: Energy expenditure and plasma F2-isoprostanes across the menstrual cycle — http://doi.org/10.1249/MSS.0b013e3181fc5eab
- See also: Psychometric characteristics of the FertiQoL questionnaire in a German sample of infertile individuals and couples — http://doi.org/10.1186/s12955-018-1058-9
- See also: Cross-cultural comparison of fertility specific quality of life in German, Hungarian and Jordanian couples attending a fertility center — http://doi.org/10.1186/s12955-016-0429-3
- See also: Detection of physical activity types using triaxial accelerometers — http://doi.org/10.1123/jpah.2011-0347